CLINICAL TRIAL: NCT00922935
Title: A 3 Arm Controlled Randomised Study: Comparison of Early and Late Loading Protocols in Full Arch Reconstructions in the Edentulous Maxilla, Using The Cresco Prosthetic System on Straumann Implants
Brief Title: Comparison of Early and Late Loading in the Edentulous Upper Jaw Using Cresco Prosthetic System on Straumann Implants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR 02/04
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Results first posted 2011-07-12 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Jaw, Edentulous
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cresco early loading (Experimental): The implants must be restored (loaded) with a permanent screw retained fixed partial denture (FPD) at 10 days of post surgery
  Interventions: Device: Cresco
- Cresco late loading (Experimental): Healing caps will be placed until loading. The minimum waiting time is 4 weeks, but not before "try ins" to ensure a perfect fit. The implants must be restored (loaded) with a permanent screw retained fixed partial denture (FPD) within 42-56 days (6 to 8 weeks) of surgery.
  Interventions: Device: Cresco
- Straumann system late loading (Active Comparator): Straumann components loading at 6-8 weeks post surgery
  Interventions: Device: Straumann components

INTERVENTIONS:
Device: Cresco — Cresco components loading 10 days post surgery
  Arms: Cresco early loading
Device: Cresco — Cresco loading at 6-8 weeks post surgery
  Arms: Cresco late loading
Device: Straumann components — Straumann components loading 6-8 weeks post surgery
  Arms: Straumann system late loading

SUMMARY:
Comparison of early and late loading of implants supporting full each prosthesis in upper jaw, using the Cresco prosthetic system on Straumann implants. The study hypothesis is that there is no difference between the bone loss (or gain) between the groups.

DETAILED DESCRIPTION:
The study is a controlled randomised study whereby each patient will receive 5-6 implants placed in the edentulous upper jaw supporting a 10-12 unit screw-retained fixed partial denture (FPD). The main objective of the study is to evaluate the performance of Straumann implants supporting a FPD using Straumann Implants and Cresco restorative components in early and delayed loading protocols at one year post-loading. The treatment groups consist of an early loading and delayed loading arm using Cresco restorative components loading time 10 days post surgery and at 6-8 weeks respectively. The control group comprise the standard delayed loading protocol (healing period 6-8 weeks) and Straumann restorative components. The primary objective is to compare changes in crestal bone levels on radiographs between implants in the control group and test groups at 1 year.The patients will be followed for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Males and females must be at least 18 years of age.
* Be edentulous in the maxilla and subjectively desire an implant supported screw retained FPD
* The teeth at the implant site must have been extracted or lost at least 3 months before the date of implantation.
* In the case of Guided Bone Regeneration(GBR) or Guided Tissue Regeneration (GTR) treatments, these procedures must have been completed at least 6 months prior to intended surgery date (to fulfil point 5).
* Adequate bone quality and quantity at the six, minimum five, implant sites to permit the insertion of Straumann 4.1 and 3.3 mm diameter implants without the use of concurrent bone augmentation techniques. I.e. implant insertion sites must have sufficient bone height such that the implant will not encroach on vital structures and sufficient width that a minimum of 1 mm of palatal and buccal bone will remain.
* Patients must be committed to participate in the study for three years follow-up examinations

Exclusion Criteria:

* Presence of conditions requiring chronic routine prophylactic use of antibiotics (e. g., history of rheumatic heart disease, bacterial endocarditis, cardiac valvular anomalies, prosthetic joint replacements)
* Medical conditions requiring prolonged use of steroids
* History of leukocyte dysfunction and deficiencies
* History of bleeding disorders
* History of neoplastic disease requiring the use of radiation or chemotherapy
* Patients with history of renal failure
* Patients with metabolic bone disorders
* History of uncontrolled endocrine disorders
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene
* Use of any investigational drug or device within the 30-day period immediately prior to implant surgery on study day 0.
* Alcoholism or drug abuse
* Patients infected with HIV
* Patients who smoke more than 10 cigarettes per day or cigar equivalents, or who chew tobacco (not greater than 10 cigarette equivalents)
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, unreliability.
* Local inflammation, including untreated periodontitis
* Mucosal diseases such as erosive lichen planus
* History of local irradiation therapy
* Presence of osseous lesions
* Unhealed extraction sites (less than 3 months post extraction of teeth in intended sites)
* Bone surgery (bone grafts, guided tissue regeneration technique for bone enhancement) at implant placement.
* Severe bruxing or clenching habits
* Persistent intraoral infection
* Patients with inadequate oral hygiene or unmotivated for adequate home care
* Lack of primary stability of 1 or more implant(s) at surgery. In this instance the patient must be withdrawn and treated accordingly.
* Insufficient bone
* Other: Inability to place implants according to protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-10; Primary Completion 2009-02 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Ellner, DDS, PhD, Principal Investigator — STP Oral protetik, Kalmar, Sweden; Asbjorn Jokstad, Professor, Principal Investigator — University of Toronto, Faculty of Denistry, 124 Edward Street, Toronto
Locations (2):
- Sweden (2):
  - STP Oral protetik, Kalmar
  - Oral rehabilitering, Linköping

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jokstad A, Ellner S, Gussgard A. Comparison of two early loading protocols in full arch reconstructions in the edentulous maxilla using the Cresco prosthetic system: a three-arm parallel group randomized-controlled trial. Clin Oral Implants Res. 2011 May;22(5):455-63. doi: 10.1111/j.1600-0501.2010.02156.x. Epub 2011 Mar 24. PMID 21435016

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cresco Early Loading | Cresco Late Loading | Straumann System Late Loading
Started | 10 | 16 | 10
Completed | 9 | 11 | 10
Not Completed | 1 | 5 | 0
Not completed — Protocol Violation | 0 | 3 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cresco Early Loading | Cresco Late Loading | Straumann System Late Loading | Total
Number analyzed (Participants) | 10 | 16 | 10 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 9 | 6 | 18
  >=65 years | 7 | 7 | 4 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (12.2) | 64.2 (10.7) | 67.1 (7) | 65.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 9 | 20
  Male | 7 | 8 | 1 | 16
Region of Enrollment [Number; unit: participants]
  Sweden | 10 | 16 | 10 | 36

OUTCOME MEASURES:

1. Primary Outcome: Bone Level Change on Radiographs
Description: Crestal bone level change at implant margin.The difference between baseline and 3 years after loading.
Time Frame: 3 years after loading
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Cresco Early Loading | Cresco Late Loading | Straumann System Late Loading
Number analyzed (Participants) | 10 | 16 | 10
mm | 2.91 (0.7) | 2.11 (0.64) | 1.70 (0.94)

ADVERSE EVENTS:
Arm/Group | Cresco Early Loading | Cresco Late Loading | Straumann System Late Loading
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/16 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/16 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cresco Early Loading (N=10) | Cresco Late Loading (N=16) | Straumann System Late Loading (N=10)
Trombosis left leg (Blood and lymphatic system disorders) | 1 (1) | 0/0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Disoriented, depressed (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — The patient came to the doctor and was depressed and disoriented. She was hospitalised and medicated and the adverse event was resolved without sequelae

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No